CLINICAL TRIAL: NCT06182839
Title: Canagliflozin in Advanced Renal Disease With MRI Endpoints
Acronym: CARe-MRI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, Thomas Mavrakanas, Assistant Professor of Medicine, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-10313
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: ESRD, CKD Stage 4, CKD Stage 5
Keywords: Canagliflozin, Advanced CKD, ESRD, Hemodialysis, Peritoneal dialysis, Cardiac MRI, SGLT-2 inhibitors
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic | interventions — Canagliflozin

STUDY DESIGN:
Intervention Model Description: We will conduct a single centre, prospective, randomized, parallel group (Canagliflozin VS placebo), double blind interventional study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be blinded to study participants and study investigators. Therefore, investigators who will interpret the cardiac magnetic resonance imaging (MRI) and who will adjudicate adverse events will be blinded to treatment group assignment. Canagliflozin 300 mg will be encapsulated to match the placebo.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Canagliflozin (Invokana) 300 mg tablet (Active Comparator)
  Interventions: Drug: Canagliflozin 300Mg Tab
- Placebo tablet (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Canagliflozin 300Mg Tab — Patients will get 1 pill of Canagliflozin 300 mg daily for one year.
  Arms: Canagliflozin (Invokana) 300 mg tablet
Drug: Placebo — Patients will get 1 pill of placebo daily for one year.
  Arms: Placebo tablet

SUMMARY:
This is a phase II, proof of concept, placebo-controlled, randomized clinical trial, assessing the effect of canagliflozin on cardiac structure and function in patients with advanced renal disease, including those on maintenance dialysis.

Our primary aim is to determine the effect of canagliflozin on cardiac structure and function in patients with advanced chronic kidney disease (CKD), compared with placebo. We hypothesize that canagliflozin will improve left ventricular (LV) hypertrophy in patients with advanced CKD. Our secondary aims are to describe the effect of canagliflozin on other cardiac magnetic resonance imaging parameters and surrogate markers of efficacy in this population.

DETAILED DESCRIPTION:
Patients with advanced renal disease, including those on maintenance dialysis, will be randomized to receive canagliflozin 300 mg orally once daily or matching placebo for one year. For patients who are not yet on renal replacement therapy, the study medication will be continued when they transition to dialysis or when they get a kidney transplant.

The prescription of all other medications, including dialysis prescription for dialysis-dependent patients, will be left to the treating physician's discretion. We will discourage changes to medications during follow-up unless deemed clinically necessary. All medications changes will be recorded at each visit.

Symptoms and adverse events will be monitored closely. Participants who experience adverse events classified as severe and probably or definitely related to the study medication will be withdrawn. Patients who develop intercurrent illnesses, are hospitalized, or have surgery (urgent or elective) will temporarily discontinue the drug.

ELIGIBILITY:
Inclusion Criteria:

* advanced CKD, defined as an estimated glomerular filtration rate (eGFR) < 20 ml/min/1.73m2 not yet on dialysis OR incident hemodialysis or peritoneal dialysis patients (i.e., who were started on dialysis in the last 6 months)*

  * For patients who were not previously followed in a CKD clinic and for whom it is not clear whether dialysis was initiated after an acute deterioration in renal function that is potentially reversible, at least 90 days of dialysis will be required prior to enrolment. This criterion only applies to patients for whom baseline eGFR prior to the acute event was ≥ 20 ml/min/1.73m2 or was unknown. The average creatinine values over the last 12 months will be used to calculate baseline eGFR.
* LV hypertrophy, defined as LV mass > 130 g/m2 in men and 100 g/m2 in females OR hospitalization for heart failure or atherosclerotic cardiovascular (CV) disease in the last 12 months OR type 2 diabetes OR UACR > 200 mg/g on a morning spot urine collection (this criterion is not applicable to patients who are on dialysis and have a urine output < 500 ml per day).

Exclusion Criteria:

* type 1 diabetes,
* history of euglycemic ketoacidosis,
* known hypersensitivity to sodium-glucose cotransporter-2 (SGLT-2) inhibitors,
* hemodynamic instability (defined as current use of parenteral inotropic agents),
* systolic BP < 90 mmHg,
* severe liver cirrhosis (Child-Pugh class C stage),
* acute hepatitis (defined as an alanine aminotransferase > 2.0 times the upper limit of normal [ULN] or total bilirubin >1.5 times the ULN),
* recurrent severe genital or urine infections,
* patients receiving digoxin, phenobarbital, phenytoin, rifampin, or ritonavir if these agents cannot be safely discontinued (due to inhibition of the P-glycoprotein mediated efflux of digoxin by canagliflozin or induction of Uridine 5'-diphospho-glucuronosyltransferase enzymes by the other agents),
* cardiac MRI-incompatible cardiac devices (cardiac pacemaker, implanted cardiac defibrillator, internal pacing wires, Swan-Ganz catheter, aneurysm clips),
* claustrophobia,
* cochlear implants,
* metallic body in the eyes,
* pregnancy or breastfeeding,
* and any other medical condition considered to be a contra-indication by the study physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular mass to volume ratio (LVMV) from baseline to 12 months, as assessed by cardiac MRI compared with placebo | 12 months
  Assessed on cardiac magnetic resonance imaging (MRI)

SECONDARY OUTCOMES:
Changes in left ventricular (LV) and atrial volumes from baseline to 12 months compared with placebo | 12 months
  Assessed on cardiac MRI
LV strain parameter changes from baseline to 12 months compared with placebo | 12 months
  Long-axis fractional shortening on cardiac MRI
Changes in myocardial edema and fibrosis from baseline to 12 months compared with placebo | 12 months
  Use of magnetic resonance imaging T2 and T1 maps, respectively (software cvi42).
Change in myocardial oxygenation reserve from baseline to 12 months compared with placebo | 12 months
  Use of oxygenation-sensitive cardiovascular magnetic resonance (OS-CMR) sequences.
Composite of major adverse cardiovascular events | 12 months
  Cardiovascular death, myocardial infarction, stroke, hospitalization for heart failure.
Death from any cause | 12 months
Progression to kidney failure (only for patients not yet on maintenance dialysis). | 12 months
  Initiation of maintenance hemodialysis, peritoneal dialysis, or renal transplantation.
Difference in distance in the 6-minute walk test at 12 months from baseline | 12 months
Difference in dyspnea score at 12 months from baseline | 12 months
  Using the 7-point Likert scale and Visual analog scale questionnaire.
Difference in quality of life at 12 months from baseline | 12 months
  Using the Kansas City Cardiomyopathy questionnaire.
Change in urine albumin to creatinine ratio (UACR) from baseline (only for patients not yet on maintenance dialysis) at 6 and 12 months | 6 months and 12 months
Change in N-terminal pro b-type natriuretic peptide (NT-proBNP) | 6 months and 12 months
Change in iron profile | 6 months and 12 months
Change in tubular injury biomarkers | 6 months and 12 months
  For patients not yet on maintenance dialysis.
Change in dose of erythropoietin-stimulating agents at 12 months from baseline | 12 months
Change in 24-hour ambulatory blood pressure at 12 months from baseline | 12 months
Composite of serious adverse events | 12 months
  Severe hyperkalemia (>6 mmol/l), acute kidney injury (≥ stage 2 using the AKIN criteria), and euglycemic ketoacidosis.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Mavrakanas, MD, Principal Investigator — Research Institute of the McGill University Health Center
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada